CLINICAL TRIAL: NCT00912730
Title: A Pilot Study of Intraoperative Gamma Camera Imaging During Sentinel Node Biopsy for Melanoma
Acronym: MEL50
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Craig L Slingluff, MD, University of Virginia - Human Immune Therapy Center
Other Study IDs: 13565
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Melanoma
Keywords: melanoma; imaging; sentinel node; biopsy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a single-institution pilot study seeking preliminary evidence of the usefulness of mobile gamma cameras in patients undergoing sentinel node biopsy for melanoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, AND
* plan to go to the operating room for sentinel node biopsy using technicium-99 labeled colloid.

Exclusion Criteria:

* under 18 years of age,
* unable to give informed consent, OR
* not planned to go to operating room for sentinel node biopsy using technicium-99 labeled colloid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma scheduled to undergo sentinel node biopsy as part of recommended clinical care, age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08

PRIMARY OUTCOMES:
Sensitivity of the Mobile gamma camera (MGC)for detection of sentinel nodes, compared to fixed gamma camera (primary)

SECONDARY OUTCOMES:
sensitivity of the MGC for detection of sentinel nodes, compared to handheld gamma probe (secondary)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States